CLINICAL TRIAL: NCT05943652
Title: Prevalence and Clinical Presentation of Functional Neurological Disorders in Patients With Movement Disorders - A Cross-sectional Study in the Movement Disorders Clinic of the Department of Neurology, Medical University of Graz
Brief Title: Observational Study on "Functional Overlay" in Patients With Movement Disorders
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 34-509 ex 21/22
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Conversion Disorder; Parkinson Disease; Tremor; Dystonia
Keywords: Accelerometry; Patient Health Questionnaire; Neuropsychology
MeSH Terms: conditions — Conversion Disorder; Parkinson Disease; Tremor; Dystonia | interventions — Neurologic Examination; Immunologic Memory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Parkinson Disease
  Interventions: Diagnostic Test: Neurological examination; Diagnostic Test: Anamnesis; Diagnostic Test: Neuropsychological testing; Diagnostic Test: Questionnaires; Diagnostic Test: Tremor recording
- Idiopathic Dystonia
  Interventions: Diagnostic Test: Neurological examination; Diagnostic Test: Anamnesis; Diagnostic Test: Neuropsychological testing; Diagnostic Test: Questionnaires; Diagnostic Test: Tremor recording
- Essential Tremor
  Interventions: Diagnostic Test: Neurological examination; Diagnostic Test: Anamnesis; Diagnostic Test: Neuropsychological testing; Diagnostic Test: Questionnaires; Diagnostic Test: Tremor recording
- Functional Neurological Disorder
  Interventions: Diagnostic Test: Neurological examination; Diagnostic Test: Anamnesis; Diagnostic Test: Neuropsychological testing; Diagnostic Test: Questionnaires; Diagnostic Test: Tremor recording
- Functional Cognitive Disorder
  Interventions: Diagnostic Test: Neurological examination; Diagnostic Test: Anamnesis; Diagnostic Test: Neuropsychological testing; Diagnostic Test: Questionnaires; Diagnostic Test: Tremor recording
- Alzheimer Disease
  Interventions: Diagnostic Test: Neurological examination; Diagnostic Test: Anamnesis; Diagnostic Test: Neuropsychological testing; Diagnostic Test: Questionnaires; Diagnostic Test: Tremor recording

INTERVENTIONS:
Diagnostic Test: Neurological examination — A neurological examination following a protocol to detect positive signs of functional neurological disorders.
Diagnostic Test: Anamnesis — A standardized question about the patient´s history. The response time is measured.
  Question: "Could you tell me about the problems with the movement disorder you are experiencing?"
Diagnostic Test: Neuropsychological testing — Neuropsychological cognitive testing including:
  * Montreal Cognitive Assessment (MOCA)
  * Rey-Osterrieth Complex Figure Test (ROCFT)
  * Wechsler Memory Scale IV
  * Comprehensive Trail Making Test (CTMT)
  * semantic and phonematic fluency tests
Diagnostic Test: Questionnaires — * Short Form 36 (SF 36)
  * Somatic Symptom Disorder - B Criteria Scale (SSD 12)
  * Patient Health Questionnaire 9 (PHQ 9)
  * Patient Health Questionnaire 15 (PHQ 15)
  * Generalized Anxiety Disorder 7 (GAD 7)
  * Fatigue Severity Scale (FSS)
  * Psychosomatic Competence Inventory (PSCI)
  * Work Ability Index (WAI)
  * Level of Personality Functioning Scale
  * Toronto Alexithymia Scale
  * Levels of Emotional Awareness Scale (short version)
  * Certainty About Mental States Questionnaire
  * Somatosensoric Amplification Scale
  * Personality Inventory for DSM-5 short version (PID5BF+M)
  * Childhood Trauma Questionnaire
  * European Quality of Life 5 Dimensions 5 Level Version (EQ5D5L)
Diagnostic Test: Tremor recording — Accelerometry following a standardized protocol, using a triaxial accelerometer transducer (Biometrics ACL300, Sensitivity 6 100 mV/G, Biometrics Ltd, UK)

SUMMARY:
The goal of this observational study is to learn about functional neurological disorders in patients with common non-functional movement disorders ("functional overlay"). The main questions it aims to answer are:

* What is the frequency of functional neurological disorders in patients with non-functional movement disorders (functional overlay)?
* What are the characteristics of functional neurological disorders in patients with non-functional movement disorders?

Participants will be examined clinically and electrophysiologically, the examinations consist of:

* a neurological examination
* neuropsychological testing
* electrophysiological tremor diagnostic
* questionnaires about psychological, biological and social risk factors

Researchers will compare patients with functional motor disorders to patients wit non-functional movement disorders to see if they differ from each other regarding the functional symptoms.

DETAILED DESCRIPTION:
Functional neurological disorders (FND) are common neurological disorders that are present in up to 16% of patients in neurological outpatient clinics. They are associated with a significant reduction in quality of life, can lead to permanent impairment, and have a poor prognosis, especially if the diagnosis is delayed.

FND have multifactorial causes and risk factors, including psychological stressors, childhood trauma, female gender, psychiatric disorders such as depression, anxiety disorder, or post-traumatic stress disorder, and other functional disorders such as irritable bowel syndrome or chronic pain syndrome. Patients with FND often report additional cognitive complaints ("cognitive fog").

A mismatch of various regulatory mechanisms, a disruption of sensory processing and motor output is assumed to be a central part of the pathogenesis. A characteristic feature of FND is a variability of symptoms according to attention. FND can be intensified by increased attention and weakened by distraction. Positive diagnostic criteria for FND have been established recently, so that by definition FND are no longer a diagnosis of exclusion.

The clinical presentations of FND are diverse and include impaired limb movement control, disturbances in vigilance that may be associated with seizures, and non-motor symptoms. FND often coincide and often coexist with pain, fatigue, sleep disorders, and cognitive disorders. Particularly non-motor functional symptoms are highly debilitating for patients.

The coincidence of "organic" neurological disorders and FND in the same patients ("functional overlay") is probably not uncommon, but has been investigated primarily in patients with Parkinson's Disease and epilepsy, so far. However, it is important to recognize FND in patients with movement disorders in order to treat them adequately and to protect them from incorrect treatment (surgery, unnecessary medication, etc.). However, the basic prerequisite for this is an exploration of the frequency and characteristics of the functional symptoms in movement disorders.

ELIGIBILITY:
Inclusion Criteria:

* Functional or non-functional movement disorder
* 18 to 80 years

Exclusion Criteria:

* Patient is not able to consent
* Patient is not able to understand / speak German fluently (questionnaires are available only in German)

Ages: 18 Years to 18 Years | Sex: All
Age Groups: Adult
Study Population: Patients with functional and non-functional movement disorders of the Movement Disorders Outpatient Clinic of the Department of Neurology, Medical University of Graz
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional neurological symptoms | on average 30 minutes
  Diagnosed by positive signs for functional neurological symptoms, as assessed in the neurological examination

SECONDARY OUTCOMES:
Duration of anamnesis | 1 to 3 minutes
  Duration in seconds of the response to the question: "Could you tell me about the problems with the movement disorder you are experiencing?"
Tremor diagnostic | up to 20 minutes
  Sum score of a electrophysiological test battery for psychogenic tremor, a scale from 0 to 10 with higher numbers indicating a higher probability for functional tremor
Subjective quality of life | 5 minutes
  European Quality of Life 5 Dimensions 5 Level Version (EQ 5D 5L), results in a 5-digit number that describes the patient's health state
Subjective health | up to 10 minutes
  Short Form 36 Questionnaire (SF-36), a 36 items questionnaires that results in 8 scales that describe the subjective health state of the patient, higher values indicating better health
Fatigue | up to 5 minutes
  Fatigue severity scale (FSS): 9 item questionnaire with a 7 point Likert scale, higher values indicating more fatigue
General anxiety | 3 minutes
  General anxiety disorder scale 7 (GAD-7): a 7 items questionnaire (0 to 21 points, higher values indicating more anxiety)
Somatic symptoms | 5 minutes
  Patient health questionnaire 15 (PHQ 15): a 15 item questionnaire (0 to 30 points, higher values indicating more somatic symptoms)
Depression | 3 minutes
  Patient health questionnaire 9 (PHQ 9): a 9 item questionnaire (0 to 27 points, higher values indicating more depressive symptoms)
Psychosomatic Competence | up to 10 minutes
  Psychosomatic Competence Inventory (PSCI): a 44 items questionnaire with a 6 point Likert scale, resulting in 6 subscales, higher values indicate higher psychosomatic competence
Work ability | 5 minutes
  Work ability index (WAI): 7 item questionnaire, 7 to 49 points, with higher values indicating better work ability
Trauma in childhood | up to 10 minutes
  Child Trauma Questionnaire (CTQ): 28 items questionnaire, 5 point Likert scale, resulting in 5 subscales with 5 to 25 points, with higher values indicating more trauma experience
Attachment styles | 5 minutes
  Experience of Close Relationships-Revised (ECR-RD 12): 12 items questionnaire with a 7 point Likert scale, resulting in 2 subscales
Alexithymia | 5 minutes
  Toronto alexithymia scale (TAS): 26 items questionnaire with a 5 point Likert scale, higher values indicating more alexithymia
Personality traits | up to 10 minutes
  The Personality Inventory for DSM-5 and ICD-11 Plus Modified (PID5BF + M): a 36 items questionnaire, with a 4 point Likert scale, resulting in 6 subscales
Personality functioning | up to 15 minutes
  Levels of personality functioning scale (LPFS): a 80 items questionnaire, with a 4 point Likert scale, resulting in 4 subscales
Executive function | up to 10 minutes
  Comprehensive trail making test (CTMT)
Memory | up to 15 minutes
  Wechsler Memory Scale
Visuospatial abilities | up to 15 minutes
  Rey-Osterrieth complex figure test
Functional cognitive symptoms | up to 60 minutes
  Incongruence in cognitive tests
Semantic word fluency | 2 minutes
  number of animals that can be listed in 2 minutes
phonematic word fluency | 2 minutes
  number of words, that start with the letter "b", that can be listed in 2 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided